CLINICAL TRIAL: NCT07324603
Title: A Randomized Controlled Trial Comparing Smartphone-Based and Face-to-Face Counseling for Chronic Tinnitus
Brief Title: Smartphone-Based vs Face-to-Face Counseling for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Beyza ASTA, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: İ04-201-23; 124S118 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Tinnitus
Keywords: Chronic tinnitus; Counseling; Smartphone-based counseling; Digital Health; Mobile Application; Patient Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face Counseling (Experimental): Participants receive structured tinnitus counseling delivered in person using a standardized educational booklet over a six-week period.
  Interventions: Behavioral: Face-to-Face Tinnitus Counseling
- Smartphone-Based Counseling (Experimental): Participants receive the same structured tinnitus counseling delivered via a mobile application with sequential modules over a six-week period.
  Interventions: Behavioral: Smartphone-Based Tinnitus Counseling

INTERVENTIONS:
Behavioral: Face-to-Face Tinnitus Counseling — Structured tinnitus counseling is delivered in person using a standardized educational booklet over a six-week period.
  Arms: Face-to-Face Counseling
Behavioral: Smartphone-Based Tinnitus Counseling — Structured tinnitus counseling is delivered via a mobile application with sequential modules over a six-week period
  Arms: Smartphone-Based Counseling

SUMMARY:
This study aims to compare the effectiveness of smartphone-based counseling and face-to-face counseling in adults with chronic tinnitus. Both interventions are based on the same structured counseling protocol and are delivered over a six-week period. The primary research question is whether smartphone-based counseling can achieve clinical outcomes comparable to those of traditional face-to-face counseling in reducing tinnitus-related impact and associated symptoms.

DETAILED DESCRIPTION:
This study is a randomized, parallel-group clinical trial designed to evaluate two counseling delivery formats for chronic tinnitus. Eligible adult participants with chronic subjective tinnitus are allocated to either smartphone-based counseling or face-to-face counseling. Both groups receive the same structured counseling content, with the delivery format being the only difference between interventions.

The counseling protocol focuses on tinnitus education, correction of maladaptive beliefs, and development of coping strategies. In the face-to-face group, counseling is delivered through scheduled in-person sessions using a structured educational booklet. In the smartphone-based group, the same content is delivered through a mobile application consisting of sequential modules, including assessment, education, coping strategies, and a clinician support feature.

Participants in both groups complete baseline assessments prior to counseling and follow-up evaluations at two and six weeks. The study is designed to examine whether smartphone-based counseling can achieve outcomes comparable to traditional face-to-face counseling when a unified counseling protocol is applied.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older

Diagnosis of chronic subjective tinnitus lasting at least 6 months

Completion of a comprehensive audiological evaluation

Ability to read and understand the study materials

Adequate cognitive function as determined by a Mini-Mental State Examination score of 25 or higher

Willingness and ability to provide written informed consent

Exclusion Criteria:

Presence of objective tinnitus

History of neurological disorders

Diagnosed major psychiatric disorders

Receipt of tinnitus-related treatment within the previous 3 months

Inability to use or access the smartphone application (for technical or device-related reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Tinnitus Impact | Baseline to 6 weeks
  Change in tinnitus impact assessed using the Tinnitus Handicap Inventory (THI).

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline to 6 weeks
  Change in depressive symptoms assessed using the Beck Depression Inventory (BDI).
Sleep Quality | Baseline to 6 weeks
  Change in sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI).
Perceived Tinnitus Severity | Baseline to 6 weeks
  Change in perceived tinnitus severity assessed using a Visual Analog Scale (VAS).
Tinnitus-Related Annoyance | Baseline to 6 weeks
  Change in tinnitus-related annoyance assessed using a Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No